CLINICAL TRIAL: NCT03559985
Title: Analgesic Effect of Paracetamol in Neuropathic Pain Patients
Brief Title: Paracetamol and Neuropathic Pain
Acronym: PAeoNy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHU-389; 2017-004505-40 (Other: 2017-004505-40)
Record Dates: First submitted 2018-05-11; First posted 2018-06-18 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Neuropathic Pain
Keywords: Paracetamol; Neuropathic pain; Analgesic effect; Pharmacogenetics; Biological parameters; Cognitivo-emotional parameters
MeSH Terms: conditions — Neuralgia | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: After a week of pre-selection (D-6 to D0), each patient will receive successively in random order each of the 2 products (paracetamol and placebo) with one wash-out period of 7 days between each administration.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Paracetamol 500 mg capsules (Doliprane® 500 mg) will remain packaged in their blister packs of origin. The necessary quantity of capsules will be packaged in a box labelled at the corresponding period (period 1 or 2).
  Lactose capsules (placebo) of the same size and colour as the Paracetamol capsules (Doliprane® 500 mg) will be bought by the CHU Pharmacy from Clermont-Ferrand. The capsules will then be blistered; the necessary quantity of capsules placebo will be packaged in the same box used for paracetamol, labelled at the time of the treatment (period 1 or 2).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol and placebo comparator (Group 1) (Other): Neuropathic pain patients taking either paracetamol or placebo according to the randomization plan
  Interventions: Drug: paracetamol; Other: Placebo comparator
- Paracetamol and placebo comparator (Group 2) (Other): Neuropathic pain patients taking either paracetamol (if during period 1 they received placebo) or placebo (if during period 1 they received paracetamol)
  Interventions: Drug: paracetamol; Other: Placebo comparator

INTERVENTIONS:
Drug: paracetamol — Period 1 (D1 to D7): 500 mg (paracetamol or placebo) to be repeated if necessary, depending on the intensity of pain, after 4 hours minimum between each treatment intake, with a maximum dose of 3 g/day, corresponding to 6 capsules per day.
  Wash-out period (D8 to D14): patients should not take paracetamol during this week.
  Period 2 (D15 to D21): 500 mg per dose (paracetamol or placebo) to be repeated if necessary, depending on the intensity of pain, after 4 hours minimum between each treatment intake, with a maximum dose of 3 g/day, corresponding to 6 capsules per day.
Other: Placebo comparator — Period 1 (D1 to D7): 500 mg (paracetamol or placebo) to be repeated if necessary, depending on the intensity of pain, after 4 hours minimum between each treatment intake, with a maximum dose of 3 g/day, corresponding to 6 capsules per day.
  Wash-out period (D8 to D14): patients should not take paracetamol during this week.
  Period 2 (D15 to D21): 500 mg per dose (paracetamol or placebo) to be repeated if necessary, depending on the intensity of pain, after 4 hours minimum between each treatment intake, with a maximum dose of 3 g/day, corresponding to 6 capsules per day.

SUMMARY:
The aim of this study is to evaluate the analgesic effect of paracetamol in patients suffering from pain with a peripheral neuropathic component in the presence of their usual treatment.

DETAILED DESCRIPTION:
This is an interventional, randomized, placebo-controlled, double-blind, crossover study about the use of paracetamol in therapeutic doses in peripheral neuropathic pain patients. The analgesic effect of paracetamol will be assessed by the painful intensity measured by numerical pain rating scale over one week after taking paracetamol/placebo.

The secondary objectives will be:

* To determine the number of patients in whom paracetamol is effective in reducing pain by at least 30% and 50%,
* To evaluate the effect of paracetamol on pain, on the number and intensity of paroxysms,
* To evaluate paracetamol consumption,
* To evaluate the effect of paracetamol on neuropathic pain patient,
* To evaluate the effect of paracetamol on mechanical allodynia,
* To monitor routine biological parameters (liver function),
* Compare Glutathione (GSH) concentrations before and after taking paracetamol,
* To perform a blood test for paracetamol and its metabolites before and after each study period,
* To perform urine dosage of paracetamol and its metabolites before and after each study period,
* To study pharmacogenetics parameters,
* To evaluate patient feeling and satisfaction after taking paracetamol,
* To evaluate the effect of paracetamol on cognition, anxiety, depression and sleep by different questionnaires,
* To collect adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 65 years,
* Patient suffering from chronic pain (for more than 3 months) with the characteristics of peripheral neuropathy and having pain assessed by a numerical scale ≥ 3 for one week, with at least 10 assessments completed,
* Patient agrees with not to take paracetamol, other than the treatment provided as part of the protocol, from inclusion to completion of the study,
* Acceptance to give a written consent.

Exclusion Criteria:

* Patient taking paracetamol daily,
* Patient with a contraindication to paracetamol administration (liver or renal failure, ...),
* Patient with a biological evaluation evaluated by the investigator as not compatible with the trial,
* Patient with a medical and/or surgical history evaluated by the investigator to be not compatible with the trial,
* Patient with drug treatments evaluated by the investigator to be not compatible with the trial,
* Pregnant or nursing woman,
* Patient with a cooperation and an understanding that does not allow for a strict compliance under the conditions set out in the protocol,
* Patient participating in another clinical trial, or being in an exclusion period, or having received a total amount of compensation exceeding 4500 euros over the 12 months preceding the start of the trial,
* Patient benefiting from a legal protection measure (curatorship, guardianship, protection of justice...),
* Patient not affiliated to the French Social Security system,
* Paracetamol intake during wash-out period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity change between period 1 and 2 | Day 1 to Day 7 (one week) and Day 15 to Day 21 (one week).
  Pain intensity change between period 1 and 2, measured by numerical pain rating scale (NPRS) over one week (two evaluations per day, morning and evening) following the taking of paracetamol/ placebo.

SECONDARY OUTCOMES:
Treatment responders at 30% (NPRS) | During 2 days before period 1 (mean of Day -1 and Day 0) and at the end of period 1 (mean of Day 6 and Day 7); during 2 days before period 2 (mean of Day 13 and Day 14) and at the end of period 2 (mean of Day 20 and Day 21).
  Calculation of the decrease of NPRS by at least 30% between the beginning and the end of the treatment period (at least 30% difference between the average of four NPRS measurements over 2 days before the start of the treatment period and the average of the four NPRS measurements over 2 days at the end of the treatment period). The number of paracetamol responders will be compared to the number of placebo responders.
Treatment responders at 50% (NPRS) | During 2 days before period 1 (mean of Day -1 and Day 0) and at the end of period 1 (mean of Day 6 and Day 7); during 2 days before period 2 (mean of Day 13 and Day 14) and at the end of period 2 (mean of Day 20 and Day 21).
  Calculation of the decrease of NPRS by at least 50% between the beginning and the end of the treatment period (at least 50% difference between the average of four NPRS measurements over 2 days before the start of the treatment period and the average of four NPRS measurements over 2 days at the end of the treatment period). The number of paracetamol responders will be compared to the number of placebo responders.
Number of paroxysms | Before period 1 (Day -6 to Day 0), over a week during period 1 (Day 1 to Day 7), over a week during wash-out (Day 8 to Day 14) and over a week during period 2 (Day 15 to Day 21).
  The number of paroxysms will be listed by the patient in the daily pain diary during all the study (28 days).
Paroxysms intensity (NPRS) | (Day -6 to Day 0), over a week during period 1 (Day 1 to Day 7), over a week during wash-out (Day 8 to Day 14) and over a week during period 2 (Day 15 to Day 21).
  The average pain of paroxyms will be evaluated by the patient in the daily pain diary during all the study (28 days). The pain intensity will be measured by NPRS: the scale ranges from 0 no pain to 10 maximal tolerable pain
Assessment of paracetamol (and placebo) consumption | At Day1, Day8, Day15, Day22
  The number of paracetamol (and placebo) capsules intake will be listed by the patient in the pain diary during the 4 weeks of the study.
Assessment of dynamic mechanical allodynia | At Day1, Day8, Day15, Day22
  Dynamic mechanical allodynia (DMA) will be evaluated by a standardized fine filament brush (Somedic, ~200-400mN) which will be moved laterally, slowly and without support, with a movement back and forth over an area of skin. Patients will be seated comfortably in a quiet room. This light touch will be applied 5 times. The sensation perceived by the patient, during each stimulus, will be rated using an ENV (0 - 10), where a score of 0 equals "no pain" and a score of 10 equals "pain maximum imaginable". The DMA will be quantified as the geometric mean of all scores corresponding to each stimulation
Assessment of liver and renal functions | At Day-6, Day1, Day8, Day15, Day22
  A tube will be taken for biochemistry analysis of alanine amino transferase, aspartate aminotransferase and bilirubin to assess the liver function and creatine level to assess the renal function at each visit. The assays will be carried out by the medical biochemistry laboratory of Clermont-Ferrand University Hospital.
Blood dosage of glutathione | At Day-6, Day1, Day8, Day15, Day22
  In order to measure the plasma glutathione level, a blood sample will be taken at each visit. After centrifugation, an aliquot will be performed to recover the plasma. The tubes will be frozen at -80°C for subsequent dosage.
Blood dosage of paracetamol and its metabolites | At Day1, Day8, Day15, Day22
  In order to determine the plasma concentration of paracetamol and its metabolites, four blood samples will be taken at D1, D8, D15 and D22. After centrifugation, an aliquot will be performed to recover the plasma. The tubes will be frozen at -80°C for subsequent dosage.
Urinary dosage of paracetamol and its metabolites | At Day1, Day7, Day15, Day21
  In order to determine the urinary concentration of paracetamol and its metabolites, four urine samples will be taken before and after each study period at D1, D7, D15 and D21 and will be frozen at -20°C for subsequent dosage.
Analysis of pharmacogenetics parameters | At the pre-selection visit (Day-6).
  Pharmacogenetics screening will focus on the metabolism of paracetamol and more specifically on the detection of the presence of one or more variant(s) of the genes UGT2B15, SULT1A1 and TRPV1. This screening will be performed on a single blood sample on D-6 (first visit). Two tubes will be taken and placed directly in the freezer at -80°C. This biological collection will be kept until the analysis.
Impact of paracetamol on patient feeling and satisfaction by Global Patient Impression of Change (PGIC) | At Day1, Day8, Day15, Day22
  This scale is used to assess patient satisfaction with treatment by choosing an answer among 8 responses (ranging from "very strongly enhanced" to "very strongly improved") to reflect their overall health.
Impact of paracetamol on cognitive parameters evaluated by Cantab® tests: Motor Screening Test (MOT), Stocking of Cambridge (SOC), Information Sampling task (IST). | At Day1, Day8, Day15, Day22
  The Cantab® test is a validated tool for exploring cognitive functions. It consists of a choice of tests that explore several cognitive dimensions: Planning (IST), Decision-making (SOC). The tests are done on a computer screen with a record of the score obtained for each test. The scores of the different tests are added and the total score compared between the 2 groups. Patients will be required to complete these tests once during their visits.
Emotional status by Hospital Anxiety and Depression scale (HAD) | At Day1, Day8, Day15, Day22
  The Hospital Anxiety and Depression scale is a self-administered questionnaire in 14 items completed by the patient. It is used to determine the levels of anxiety and depression. Seven of the items relate to anxiety and seven relate to depression. Global score ranges from 0 to 42.
Sleep by the Pittsburgh Sleep Quality Index (PSQI) | At Day1, Day8, Day15, Day22
  This questionnaire consists of 19 items and is used to measure sleep quality. It consists of 7 domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction.
Descriptive analysis of adverse event of paracetamol use. | Pain diary: over 4 weeks: At the pre-selection visit (Day -6) to the end of the study (Day 22).
  The adverse event will be reported by the patient on his pain diary during all the study. Furthermore, a daily phone-call will be performed by the team project during the two period of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Lise LACLAUTRE, Clermont-Ferrand, France